CLINICAL TRIAL: NCT00496964
Title: Botox for Non-surgical Lateral Release in Patellofemoral Pain
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Insufficient recruitment in a reasonable time + expiration of study medication
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PT_PMR_3700
Record Dates: First submitted 2007-07-05; First posted 2007-07-06 (Estimated); Results first posted 2011-05-18 (Estimated); Last update posted 2017-10-23 (Actual); Status verified 2017-09

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: Botulinum toxin type A; Patellofemoral pain syndrome; Knee Injuries; Exercise Therapy
MeSH Terms: conditions — Patellofemoral Pain Syndrome; Knee Injuries | interventions — Botulinum Toxins, Type A; Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Injection of Botulinum toxin A into vastus lateralis of study limb plus exercise program
  Interventions: Drug: Botulinum toxin A + exercise
- 2 (Placebo Comparator): Placebo injection + exercise
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Botulinum toxin A + exercise — Injection of 100 units Botox (Botulinum toxin type A) into the Vastus Lateralis of the study leg + 12 weeks of exercise for patellofemoral pain
  Other Names: Botox
  Arms: 1
Drug: Placebo — Injection of 2 cc placebo containing 0.1cc sodium bicarbonate 8.4% (1meq/cc), 0.9cc normal saline and 1 cc of lidocaine into the vastus lateralis of the study leg followed by 12 weeks of exercise for patellofemoral pain syndrome
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether the use of botulinum toxin A injected into the lateral thigh muscle improves knee function and reduces knee pain secondary to patellofemoral syndrome. The study hypothesis is that botulinum toxin + specific exercises will be superior to specific exercises alone in improving knee function and reducing knee pain in individuals with patellofemoral syndrome.

DETAILED DESCRIPTION:
Patellofemoral pain syndrome is a leading cause of knee pain in persons under 45 and is particularly common in women. The prevailing theory for the etiology of patellofemoral pain is an imbalance in force or timing of the pull of the knee extensor muscles on the patella resulting in improper tracking of the patella in the femoral grove. Specifically, the vastus medialis is thought to be ineffective in overcoming the lateral pull of the vastus lateralis. When exercises designed to focus on improving strength and timing of activation of the vastus medialis fail, surgical release of part of the attachment of the vastus lateralis to the patella is considered.

Botulinum toxin temporarily blocks acetylcholine release from motor neurons and is used clinically to produce muscle relaxation.

Subjects with patellofemoral syndrome will be recruited into the study. Half of the subjects will be given a placebo injection while the other half will be given an injection of Botox (Botulinum Toxin A, Allergen) into the vastus lateralis muscle. Group assignment will be randomized and a double blind protocol used. Prior to injection, the subject will record their level of knee pain, fill out several knee function questionnaires, and have the strength and endurance of their knee extensor muscles tested. All subjects will be given an exercise program designed to target strengthening of the medial thigh muscles as well as stretching of lateral structures.

At 4, 6 and 12 weeks knee pain and knee function will again be assessed.

ELIGIBILITY:
Inclusion Criteria:

* retropatellar knee pain
* pain with two of: prolonged sitting, climbing stairs, squatting, running, kneeling, hopping, jumping
* pain with patellar palpation
* symptoms minimum 1 month
* Visual Analog Scale for pain (VAS) usual pain 4 of 10 on VAS [0-10 scale, anchors 0 = no pain, 10 = worst pain imaginable]

Exclusion Criteria:

* history knee surgery
* history patellar dislocation
* clinical evidence of meniscal lesion, ligamentous instability, traction apophysitis around the patellofemoral complex, patellar tendon pathology, chondral damage, osteoarthrosis, spinal referred pain

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2005-05; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sheryl D Finucane, PhD, PT, Principal Investigator — Department of Physical Therapy, Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

REFERENCES:
- [Background] Singer BJ, Silbert PL, Dunne JW, Song S, Singer KP. An open label pilot investigation of the efficacy of Botulinum toxin type A [Dysport] injection in the rehabilitation of chronic anterior knee pain. Disabil Rehabil. 2006 Jun 15;28(11):707-13. doi: 10.1080/09638280500301477. PMID 16809213
- [Background] Crossley K, Bennell K, Green S, McConnell J. A systematic review of physical interventions for patellofemoral pain syndrome. Clin J Sport Med. 2001 Apr;11(2):103-10. doi: 10.1097/00042752-200104000-00007. PMID 11403109
- [Background] Crossley KM, Bennell KL, Cowan SM, Green S. Analysis of outcome measures for persons with patellofemoral pain: which are reliable and valid? Arch Phys Med Rehabil. 2004 May;85(5):815-22. doi: 10.1016/s0003-9993(03)00613-0. PMID 15129407

RESULTS

PARTICIPANT FLOW:
Groups:
- Botulinum Toxin A Injection + Exercise: Injection of Botulinum toxin A into vastus lateralis of study limb plus exercise program
- Placebo Injection + Exercise: Placebo injection into Vastus Lateralis + exercise
Period: Overall Study
Arm/Group | Botulinum Toxin A Injection + Exercise | Placebo Injection + Exercise
Started | 1 | 4
Completed | 1 | 3
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Botulinum Toxin A Injection + Exercise | Placebo Injection + Exercise | Total
Number analyzed (Participants) | 1 | 4 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 4 | 5
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 | 25.5 (2.53) | 27.0 (2.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale Pain Ratings (VAS)
Description: Visual Analog Scale pain rating (VAS). 10 cm line with anchors at 0 (no pain) and 10 cm (worst imaginable pain). Scores are in cm (0 - 10) 0 no pain, higher values greater pain. Results given are for change at 12 weeks compared to baseline (week 12 score - baseline score)
Time Frame: 4, 6, 12 weeks
Population: analysis per protocol. Drop out not included in analysis. mean reduction in Visual Analog Scale for Pain (VAS) from start to 12 weeks.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Botulinum Toxin A Injection + Exercise | Placebo Injection + Exercise
Number analyzed (Participants) | 1 | 3
cm | 6 | 3.7 (0.33)

2. Primary Outcome: Change in Anterior Knee Pain Scale.
Description: Anterior Knee Pain Scale: a 13-item questionnaire; a TOTAL score of 0 = severe disability; a score of 100 = no pain or disability. (items are scored 0-5 or 0-10).
  Change scores at 12 wks are reported. Inverted so positive values reflect improvement.
  Included items: difficulty with: weight bearing, walking, stairs, squat, run, jump, prolonged sitting; presence of limp, swelling, patellar subluxation, atrophy of thigh, reduced knee flexion. Reference: Kujala et al: Scoring of Patellofemoral Disorders. J Arthroscopic Rel Surg, 9(2)159-163, 1993
Time Frame: 4, 6, 12 weeks
Population: The Anterior Knee Pain Scale is a 13-item questionnaire; a score of 0 = severe disability; a score of 100 = no pain or disability. Change scores are reported. Positive values = improvement in symptoms.
Measure: Mean (Standard Deviation); unit: Units on Scale
Arm/Group | Botulinum Toxin A Injection + Exercise | Placebo Injection + Exercise
Number analyzed (Participants) | 1 | 3
Units on Scale | 19 | 16.7 (4.37)

3. Primary Outcome: Functional Index Questionnaire
Description: The Functional Index Questionnaire (FIQ) is a self report functional rating scale. Individuals rate eight-activities. Each activity is rated from 0 - 2 with ) being unable to perform the activity and 2 being able to perform the activity without difficulty. The total score is summed for a final score of 0 - 16. 0 indicates that the individual is ubable to perform any of the tasks, 16 indicates that the subject is able to perform all tasks without difficulty. The eight items include: walking (1 block and 1 mile), climbing stairs (2 flights and 4 flights), squatting, kneeling, prolonged sitting, and running
Time Frame: 4, 6, 12 weeks
Population: No statistical analysis due to small number of subjects
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Botulinum Toxin A Injection + Exercise | Placebo Injection + Exercise
Number analyzed (Participants) | 1 | 3
units on a scale
  Pre | 11 (NA) — only one subject | 10 (1.7)
  Post 4 wk | 12 (NA) — only one subject | 10 (1.7)
  Post 6 wk | 11 (NA) — only one subject | 10.7 (0.6)
  Post 12 wk | 13 (NA) — only one subject | 14 (1.7)

4. Primary Outcome: Lower Extremity Functional Scale
Description: The lower extremity functional scale (LEFS) is a self report questionnaire. Subjects rate 19 items related to general activities that require the lower extremities on a scale of 0 - 4. 0 = extreme difficulty or unable to perform the activity, 4 = No difficulty performing the activity. The total of all rankings are summed and divided by the maximum score (76). The score is reported as a percentage. 100% = no difficulty in performing any of the tasks. 0% = extreme difficulty or unable to perform all of the tasks.
Time Frame: 4, 6, 12 weeks
Population: No statistical analysis due to small number of subjects
Measure: Mean (Standard Deviation); unit: percentage of total possible score
Groups:
- Botulinum Toxin A Injection + Exercise: Subjects in this group received an Injection of Botulinum toxin A in the vastus lateralis of the study limb plus exercise program
  Subjects received a single injection of 100 ml of Botulinum toxin A (Botulinum toxin type A) into the vastus lateralis muscle of the involved limb near the motor point followed by instruction in a home exercise program for knee and hip musculature that Exercises were performed for 12 weeks, with the number or repetitions and sets determined and progressed by a physical therapist based on reports of knee pain.
- Placebo Injection + Exercise: Placebo injection + exercise
  Placebo: Injection of 2 cc placebo containing 0.1cc sodium bicarbonate 8.4% (1meq/cc), 0.9cc normal saline and 1 cc of lidocaine into the vastus lateralis of the study leg followed by 12 weeks of exercise for patellofemoral pain syndrome focusing on the knee & hip.
Arm/Group | Botulinum Toxin A Injection + Exercise | Placebo Injection + Exercise
Number analyzed (Participants) | 1 | 3
percentage of total possible score
  Pre | 69 (NA) — only one subject | 66.7 (14.6)
  Post 4 wks | 87 (NA) — only one subject | 71 (8)
  Post 6 wks | 87 (NA) — only one subject | 73 (11.4)
  Post 12 wks | 91 (NA) — only one subject | 75 (14)

5. Secondary Outcome: Maximal Knee Extensor Force During Concentric and Isometric Contractions
Time Frame: 4, 6, 12 weeks
Measure: Mean (Standard Deviation); unit: Nm
Arm/Group | Botulinum Toxin A Injection + Exercise | Placebo Injection + Exercise
Number analyzed (Participants) | 1 | 3
Nm
  Isometric Torque 30deg pre | 26 (NA) — only one subject | 31.3 (13.1)
  Isometric Torque 30deg 4w | 57 (NA) — only one subject | 43.7 (8.1)
  Isometric Torque 30deg 6w | 43 (NA) — only one subject | 39.0 (2.65)
  Isometric Torque 30deg 12w | 37 (NA) — only one subject | 42.3 (5.1)

6. Secondary Outcome: Knee Extensor Fatigue
Description: This is not available due to data collection errors
Time Frame: 4, 6, 12 weeks
Population: This is not available due to data collection errors
Arm/Group | Botulinum Toxin A Injection + Exercise | Placebo Injection + Exercise
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Muscle Activation During Maximal Contractions and Fatigue Contractions
Description: muscle activation as EMG ratios of VMO/VL at 30 degrees maximal isometric contraction at 30degrees
Time Frame: 4, 6, 12 weeks
Measure: Mean (Standard Deviation); unit: ratio VMO EMG to VL EMG
Arm/Group | Botulinum Toxin A Injection + Exercise | Placebo Injection + Exercise
Number analyzed (Participants) | 1 | 3
ratio VMO EMG to VL EMG
  EMG ratio VMO/VL pre | 0.91 (NA) — Only one subject | 0.6 (0.14)
  EMG ratio VMO/VL 4wk | NA (NA) — Equipment error during data collection session resulted in invalid data | 0.61 (0.35)
  EMG ratio VMO/VL 6wk | 0.54 (NA) — Only one subject | 0.50 (0.15)
  EMG ratio VMO/VL 12wk | 0.55 (NA) — Only one subject | 0.69 (0.33)

ADVERSE EVENTS:
Arm/Group | Botulinum Toxin A Injection + Exercise | Placebo Injection + Exercise
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/4
Other Adverse Events (participants affected / at risk) | 0/1 | 0/4

LIMITATIONS AND CAVEATS:
Early termination due to small number of subjects. No statistical analysis of data due to small number of subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No